CLINICAL TRIAL: NCT03417908
Title: Effects of Proprioceptive Neuromuscular Facilitation Applied to the Accessory Respiratory Muscles on Functional and Electromyographic Parameters in Patients With and Without COPD
Brief Title: Respiratory Muscle Stretching Effect on Functional and Electromyographic Parameters of Patients With and Without COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Pampa (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Anelise Dumke, Professor, Universidade Federal do Pampa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-411
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-02

CONDITIONS: COPD
Keywords: Proprioceptive neuromuscular facilitation; Pulmonary Rehabilitation; muscle activation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD - PNF (Active Comparator): COPD - PNF
  Interventions: Procedure: PNF
- COPD - sham (Sham Comparator): COPD - sham
  Interventions: Procedure: Sham
- Individuals Without COPD - PNF (Active Comparator): Individuals Without COPD - PNF
  Interventions: Procedure: PNF
- Individuals Without COPD - sham (Sham Comparator): Individuals Without COPD - sham
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: PNF — The contract-relax method of proprioceptive neuromuscular facilitation (PNF) technique will be used for stretching of ESC, ECM and external intercostals muscles. The contraction of agonist muscles against the resistance imposed by the physiotherapist (isometric contraction) will be maintained for 6 seconds. After that, the patient is oriented to relax the muscles for 6 seconds without losing range of motion, and then the muscle will be lengthened. This procedure is repeated until the maximum amplitude of motion of the neck and upper limb is reached. The stretching will be performed on the right and left sides of the body.
  Arms: COPD - PNF; Individuals Without COPD - PNF
Procedure: Sham — Isotonic concentric contraction of the biceps (two sets of five push-ups elbow in both arms) with the individual sitting in a chair with back support.
  Arms: COPD - sham; Individuals Without COPD - sham

SUMMARY:
To evaluate the activation of accessory respiratory muscles and the effects of stretching these muscles in patients with COPD.

DETAILED DESCRIPTION:
All subjects (sixty men) will perform spirometry, measure of inspiratory capacity (IC) and maximal inspiratory and expiratory pressures (MIP and MEP). Baseline blood pressure (BP), respiratory rate (RR), heart rate (HR), sensation of dyspnea (Borg Scale) and oxygen saturation (pulse oximetry, SpO2) will be collected prior to the performance of pulmonary function tests.

The electrical activity of the scalene (ESC), sternocleidomastoid (SCM) and external intercostal muscles (INTER) will be measured by surface electromyography (sEMG) at rest and during the maneuvers of IC, MIP and MEP.

Control group: The control group will perform isotonic concentric contraction of the biceps (two sets of five push-ups elbow in both arms) with the individual sitting in a chair with back support.

Intervention group: The contract-relax method of proprioceptive neuromuscular facilitation (PNF) technique will be used for stretching of ESC, ECM and external intercostals muscles. The contraction of agonist muscles against the resistance imposed by the physiotherapist (isometric contraction) is maintained for 6 seconds. After that, the patient will be asked to relax the muscles for 6 seconds without losing range of motion, and then the muscle will be lengthened. This procedure is repeated until the maximum amplitude of motion of the neck and upper limb is reached. The stretching will be performed on the right and left sides of the body.

Statistical analysis will be carried out with the Statistical Package for the Social Sciences, version 18.0 (SPSS Inc., Chicago, IL, USA). Normality of data distribution will be assessed by the Shapiro-Wilk test.

Values will be presented as mean ± standard deviation (SD) or median (25-75%). To compare the differences between the baseline characteristics between the groups the t test for independent samples will be used. The effect of the intervention will be evaluated by paired t test. For the analysis of the electromyographic signal will be use the Wilcoxon T test. Statistical significance is accepted at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Control group: Men without respiratory symptoms and lung disease, with normal spirometry.
* Interventional group: Men diagnosed with severe to very severe COPD (forced expiratory volume in one second / forced vital capacity - FEV1/FVC <0.7 and FEV1 <50% predicted after bronchodilator use); clinically stable over the past 4 weeks.

Exclusion Criteria:

* History of fracture in the spine and / or upper limb
* Herniated disc
* Connective tissue disease
* Ischemic heart disease or uncontrolled hypertension
* Obesity (BMI> 30 kg/m2)
* Aortic aneurysm
* Recent abdominal or thoracic surgery
* Glaucoma
* Retinal detachment

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-12-14 (Estimated); Study Completion 2018-12-14 (Estimated)

PRIMARY OUTCOMES:
Change in inspiratory capacity | One day
  Change in inspiratory capacity

SECONDARY OUTCOMES:
Change in maximal respiratory pressure (MIP and MEP) | One day
  Change in maximal respiratory pressure (MIP and MEP)
Change in electromyographic activity of accessory respiratory muscles | One Day
  Change in electromyographic activity of accessory respiratory muscles

CONTACTS AND LOCATIONS:
Overall Officials: Anelise Dumke, Principal Investigator — Federal University of Rio Grande do Sul; Marli M. Knorst, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Anelise Dumke, Uruguaiana, Rio Grande do Sul, Brazil